CLINICAL TRIAL: NCT04501718
Title: A Single Arm Clinical Phase Ⅱ Study of Apatinib Combined with Temozolomide and Etoposide Capsules in the Treatment of Recurrent Medulloblastoma in Children
Brief Title: Apatinib Combined with Temozolomide and Etoposide Capsules in the Treatment of Recurrent Medulloblastoma in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Junping Zhang, professor, Beijing Sanbo Brain Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BJ-MB-II-001
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — Temozolomide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test group (Experimental)
  Interventions: Drug: Apatinib Combined With Temozolomide and Etoposide Capsules

INTERVENTIONS:
Drug: Apatinib Combined With Temozolomide and Etoposide Capsules — Apatinib mesylate tablets: Oral, 250mg, qd. Take the medicine with warm water half an hour after a meal (the daily medicine should be taken at the same time as possible).
  28 days is a cycle, and the medication is administered until the disease progresses (PD), intolerable toxicity occurs or the patient withdraws informed consent. The longest period does not exceed 12 cycles. The treatment after 12 cycles is determined by the investigator.

SUMMARY:
This study is a prospective single-center clinical study, which aims to observe and evaluate the efficacy and safety of apatinib combined with temozolomide and oral etoposide in the treatment of recurrent medulloblastoma in children.

DETAILED DESCRIPTION:
This research plan is implemented in accordance with GCP principles in Sanbo Brain Hospital of Capital Medical University.

Subjects are screened into the group. If the following conditions do not occur (the subject withdraws the informed consent, the drug side effects are intolerable, the investigator thinks it is not suitable for further testing, etc.), the expected research treatment for each subject It will continue until tumor progression or death confirmed by imaging studies, but not more than 2 years. Observe the effectiveness index and safety index during the test.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2-21 (at the time of diagnosis), no gender limit.
2. After biopsy or surgery, the first postoperative pathological diagnosis is medulloblastoma.
3. The recurrence of the tumor is confirmed by MRI, that is, the diameter of the lesion on the enhanced MRI image is ≥1cm, and ≥2 slices (slice spacing 5mm) are visible; or after another biopsy or surgery, the pathological diagnosis is medulloblastoma.
4. The time interval from the last radiotherapy is ≥4 weeks.
5. The time interval from the last chemotherapy is ≥4 weeks, and the patients have fully recovered from the acute toxicity of the last treatment. If you receive nitrosourea chemotherapeutics before enrollment, the interval between enrollment and the last chemotherapy is ≥6 weeks.
6. The interval between the last biopsy or surgery is ≥2 weeks.
7. KPS score ≥50 (patient> 12 years old), or Lansky score ≥ 50 (patient ≤ 12 years old).
8. If the patient is taking glucocorticoid therapy, the hormone dosage has stabilized or decreased for at least 1 week before the baseline MRI.
9. The expected survival time is ≥12 weeks.
10. The main organ functions are normal, and there is no serious blood, heart, lung, liver, kidney dysfunction and immune deficiency diseases. The laboratory inspection meets the following requirements:

(1) Routine blood examination, which must be met (no blood transfusion within 14 days):

1. HGB≥100g/L;
2. WBC≥3.0×109/L; NEUT≥1.5×109/L;
3. PLT ≥100×109/L; (2) The biochemical inspection shall meet the following standards:

a. BIL≤1.5 times the upper limit of normal (ULN); b. ALT and AST≤2.0×ULN; c. Serum Cr≤1.5×ULN or endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula); (3) Occult blood in stool (-); (4) Urine routine is normal, or urine protein <(++), or 24-hour urine protein <1.0 g; 11. The ECG shows that the heart rate is in the normal range (55-100 beats/min), the QT interval is normal or slightly prolonged (QTc<480ms), the T wave is normal or low, and the ST segment is normal or non-specific changes.

12. The coagulation function is normal, without active bleeding and thrombosis.

1. International standardized ratio INR≤1.5×ULN;
2. Partial thromboplastin time APTT≤1.5×ULN;
3. Prothrombin time PT≤1.5ULN. 13. Female patients of childbearing age must undergo a negative pregnancy test (serum or urine) within 7 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 8 weeks after the last administration; male patients of childbearing age should agree to During the observation period and within 8 weeks after the last administration, use appropriate methods of contraception.

   14. Patients voluntarily provide 25-30 slices of tumor tissue after the last biopsy or surgery.

   15. The patient has normal swallowing function and can swallow capsules. 16. The patient voluntarily joined the study and signed an informed consent form (ICF).

   17. Those who are expected to have good compliance can follow up the efficacy and adverse reactions as required by the plan.

   Exclusion Criteria:
   1. Past application of anti-tumor angiogenesis drugs;
   2. Those who are known to be allergic to any component of temozolomide, apatinib, and etoposide;
   3. Are using antiepileptic drugs that induce liver drug enzymes, unless they have been replaced with antiepileptic drugs that are non-hepatic drug enzymes at least 2 weeks away from enrollment;
   4. Patients with other malignant tumors, unless they have survived without progression for 5 years and the researcher believes that the risk of recurrence is low or patients with carcinoma in situ;
   5. People with hypertension who cannot be reduced to the normal range after treatment with antihypertensive drugs (systolic blood pressure ≤140 mmHg / diastolic blood pressure ≤ 90 mmHg);
   6. Suffering from severe cardiovascular disease; T wave inverted or high tip of ECG, ST segment specific changes.
   7. Urine routine test indicates urine protein ≥(++), or 24-hour urine protein ≥1.0g;
   8. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5×ULN), have bleeding tendency or are receiving thrombolytic or anticoagulant therapy;
   9. There are many factors that affect the absorption of oral drugs, such as uncontrollable nausea and vomiting, chronic diarrhea and intestinal obstruction;
   10. There is an infection that is difficult to control;
   11. Have had significant clinically significant bleeding symptoms or a clear bleeding tendency within 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, gastrointestinal perforation, fecal occult blood++ and above at baseline, intratumoral or Intracranial hemorrhage, or suffering from vasculitis, etc.;
   12. Arterial/venous thrombosis events that occurred within 6 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
   13. Pregnant or breast-feeding women; fertility patients who are unwilling or unable to take effective contraceptive measures;
   14. Other situations that the researcher thinks are not suitable for inclusion.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 4 years
Progression-free survival (PFS) | up to 4 years
Overall survival (OS) | up to 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sanbo Brain Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No